CLINICAL TRIAL: NCT07222267
Title: A Phase 1a/1b Study Evaluating the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Preliminary Antitumor Activity of BG-75202, Alone and in Combination With Other Agents in Patients With Advanced Solid Tumors
Brief Title: An Investigational Study of BG-75202 Alone and in Combination With Other Therapeutic Agents in Adults With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: BeOne Medicines (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BG-75202-101; 2025-523553-34-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-28; First posted 2025-10-29 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer; Advanced Solid Tumor
Keywords: KAT6 inhibitor
MeSH Terms: conditions — Breast Neoplasms | interventions — Cyclin-Dependent Kinase Inhibitor p16; Estrogen Receptor Antagonists; Aromatase Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part 1A: Dose Escalation and Safety Expansion, BG-75202 Monotherapy (Experimental): Sequential cohorts of increasing dose levels of BG-75202 will be evaluated as monotherapy.
  Interventions: Drug: BG-75202
- Part 1B: Dose Escalation and Safety Expansion, BG-75202 + Estrogen Receptor Antagonist (Experimental): Sequential cohorts of increasing dose levels of BG-75202 will be evaluated in combination with an estrogen receptor antagonist.
  Interventions: Drug: BG-75202; Drug: Estrogen Receptor Antagonist
- Part 2A: Dose Optimization, BG-75202 + Estrogen Receptor Antagonist (Experimental): Participants will receive BG-75202 in combination with an estrogen receptor antagonist.
  Interventions: Drug: BG-75202; Drug: Estrogen Receptor Antagonist
- Part 2B: Safety Run-In, BG-75202 + CDK4 inhibitor + Aromatase Inhibitor (Experimental): Participants will receive BG-75202 in combination with a cyclin-dependent kinase 4 (CDK4) inhibitor and an aromatase inhibitor.
  Interventions: Drug: BG-75202; Drug: CDK4 Inhibitor; Drug: Aromatase Inhibitor
- Part 2C: Dose Expansion, BG-75202 + CDK4 inhibitor + Aromatase Inhibitor (Experimental): Participants will receive BG-75202 in combination with a CDK4 inhibitor and an aromatase inhibitor.
  Interventions: Drug: BG-75202; Drug: CDK4 Inhibitor; Drug: Aromatase Inhibitor

INTERVENTIONS:
Drug: BG-75202 — Administered orally.
Drug: CDK4 Inhibitor — Administered orally.
  Arms: Part 2B: Safety Run-In, BG-75202 + CDK4 inhibitor + Aromatase Inhibitor; Part 2C: Dose Expansion, BG-75202 + CDK4 inhibitor + Aromatase Inhibitor
Drug: Estrogen Receptor Antagonist — Administered by intramuscular injection.
  Arms: Part 1B: Dose Escalation and Safety Expansion, BG-75202 + Estrogen Receptor Antagonist; Part 2A: Dose Optimization, BG-75202 + Estrogen Receptor Antagonist
Drug: Aromatase Inhibitor — Administered orally.
  Arms: Part 2B: Safety Run-In, BG-75202 + CDK4 inhibitor + Aromatase Inhibitor; Part 2C: Dose Expansion, BG-75202 + CDK4 inhibitor + Aromatase Inhibitor

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics, and preliminary antitumor activity of BG-75202 (KAT6A/B inhibitor) alone and in combination with other therapies in participants with breast cancer and other advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Part 1A: Participants with histologically or cytologically confirmed advanced, metastatic breast cancer and other solid tumors who have exhausted, are intolerant of all available standard of care therapies, and/or without available standard of care therapies.
* Part 1B and Part 2A: Participants with advanced breast cancer with 1 to 3 prior lines of systemic therapy in the metastatic setting. Prior lines in the advanced/ metastatic setting may not exceed 2 lines of chemotherapy (inclusive of antibody-drug conjugate with cytotoxic payload).
* Parts 2B and 2C: Participants with advanced breast cancer enrolled in regions where cyclin-dependent kinase 4/6 (CDK4/6) inhibitors are not approved and/or not available as the first-line treatment and who are CDK4/6 inhibitor treatment naïve and did not receive any previous systemic treatment for advanced disease.
* Participants with breast cancer must have histologically or cytologically confirmed advanced breast cancer at the time of most recent testing, based on American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines.
* Female participants with metastatic breast cancer must be postmenopausal or receiving ovarian function suppression treatment.
* Measurable disease as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1.
* Stable Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Adequate organ function.

Exclusion Criteria:

* Prior exposure to KAT6A/B or KAT7 inhibitors/degraders.
* Patients with active leptomeningeal disease or uncontrolled, untreated brain metastasis.
* Participants with any malignancy ≤ 3 years before screening for the study except for the specific cancer under investigation in this study and any locally recurring cancer that has been treated curatively which in the opinion of the investigator is unlikely to require intervention during the study.

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-12-11 (Actual); Primary Completion 2029-04-30 (Estimated); Study Completion 2036-07-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Number of Participants with Adverse Events (AEs) | From first dose to 30 days after last dose or initiation of a new anticancer therapy, whichever occurs first, up to approximately 12 months
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including physical examination findings, electrocardiogram results, laboratory values, and AEs meeting protocol-defined dose-limiting toxicity (DLT) criteria.
Part 1: Recommended Dose for Expansion (RDFE) | Estimated approximately 1 year
  The RDFE is based on the maximum tolerated dose (MTD) or maximum administered dose (MAD) with consideration of the tolerability, pharmacokinetics (PK), pharmacodynamics, antitumor activity, and any other available relevant data.
Part 2: Overall Response Rate (ORR) | Up to approximately 2 years
  ORR is defined as the percentage of participants with partial or complete response, as assessed by the investigator using Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).

SECONDARY OUTCOMES:
Part 1: ORR | Up to approximately 1 year
  ORR is defined as the percentage of participants with partial response (PR) or complete response (CR), as assessed by the investigator using RECIST v1.1.
Part 1: Duration of Response (DOR) | Up to approximately 1 year
  DOR is defined as the time from the first determination of an objective response to disease progression documented after treatment initiation or death, whichever occurs first.
Part 1: Time to Response (TTR) | Up to approximately 1 year
  TTR is defined as the time from treatment initiation to the first determination of objective response.
Part 2: DOR | Up to approximately 2 years
  DOR is defined as the time from the first determination of an objective response to disease progression documented after treatment initiation or death, whichever occurs first.
Part 2: TTR | Up to approximately 2 years
  TTR is defined as the time from treatment initiation to the first determination of objective response.
Part 2: Disease Control Rate (DCR) | Up to approximately 2 years
  DCR is defined as the percentage of participants who achieve CR, PR, or stable disease as assessed by investigator's review.
Part 2: Clinical Benefit Rate (CBR) | Up to approximately 2 years
  CBR is defined as the percentage of participants who achieve CR, PR, or durable stable disease (stable disease ≥ 24 weeks).
Part 2: Progression-Free Survival (PFS) | Up to approximately 2 years
  PFS is defined as the time from the date of the first dose of study treatment(s) to the date of the first documentation of disease progression assessed by investigator's review or death, whichever occurs first.
Part 2: Number of Participants with Adverse Events (AEs) | Up to approximately 2 years
  Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), including physical examination findings, electrocardiogram results, and laboratory values.
Part 2: Recommended Phase 2 Dose (RP2D) | Up to approximately 2 years
  The RP2D of BG-75202 will take into consideration the totality of data including, but not limited to, PK, pharmacodynamics, safety, tolerability, and antitumor activity.
Parts 1 and 2: Maximum Observed Plasma Concentration (Cmax) of BG-75202 | Up to approximately 4 months
Parts 1 and 2: Minimum Observed Plasma Concentration (Ctrough) of BG-75202 | Up to approximately 4 months
Parts 1 and 2: Area Under the Plasma Concentration-Time Curve (AUC) of BG-75202 | Up to approximately 4 months
Parts 1 and 2: Terminal Half-Life (t1/2) of BG-75202 | Up to approximately 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — BeOne Medicines
Locations (5):
- United States (2):
  - Next Oncology Austin, Austin, Texas
  - The University of Texas Md Anderson Cancer Center, Houston, Texas
- Australia (2):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Cancer Research South Australia, Adelaide, South Australia
- Fudan University Shanghai Cancer Centerpudong, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
BeOne shares data on completed studies responsibly and provides qualified scientific and medical researchers access to data and supporting documentation for clinical trials in dossiers for medicines and indications after submission and approval in the United States, China, and Europe. Clinical trials supporting subsequent local approvals, new indications, or combination products are eligible for sharing once corresponding regulatory approvals are achieved.
  BeOne shares data only when permitted by applicable data privacy and security laws and regulations, when it is feasible to do so without compromising the privacy of study participants, and other considerations.
  Qualified researchers with appropriate competencies who are engaged in novel scientific research may submit a request for participant-level data with a research proposal for BeOne review. Research teams must include a biostatistician and sign a Data Sharing Agreement prior to receiving access to clinical trial data.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See plan description
Access Criteria: See plan description
URL: https://beonemedicines.com/science/clinical-trials/